CLINICAL TRIAL: NCT06514963
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics and Food Effect on the Pharmacokinetics of HRS-9813 Tablets After Single and Multiple Ascending Oral Doses in Healthy Volunteers
Brief Title: A Trial of HRS-9813 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-9813-101
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: HRS-9813 compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single ascending dose (SAD) cohorts (Experimental): Subjects will be assigned to one of 5 planned dose cohorts and receive single dose of HRS-9813 or placebo
  Interventions: Drug: HRS-9813; Drug: Placebo
- multiple ascending dose (MAD) cohorts (Experimental): Subjects will be assigned to one of 3-4 planned dose cohorts and receive multiple doses of HRS-9813 or placebo
  Interventions: Drug: HRS-9813; Drug: Placebo

INTERVENTIONS:
Drug: HRS-9813 — Specified dose on specified days
Drug: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this phase Ⅰ study is to evaluate the safety, tolerability and pharmacokinetics of HRS-9813 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and methods, voluntarily participate in the study, comply with study requirements, and sign the written informed consent form (ICF);
2. Male or female aged 18-55 (adult healthy volunteers);
3. Body mass index (BMI) between 19 and 26 kg/m2;
4. Normal Electrocardiogram (ECG);
5. Men and women of childbearing potential must agree to take effective contraceptive methods.

Exclusion Criteria:

1. Any significant acute or chronic medical condition that presents a potential risk to the participant and/or that may compromise the objectives of the study, including active, or history of, urinary stones, urinary tract infection, or intestinal disorder including irritable bowel syndrome;
2. History or presence of malignancy; participants with a history of basal cell or squamous cell carcinoma that has been treated with no evidence of recurrence within 5 years will be allowed for inclusion;
3. Seated systolic blood pressure (SBP) of <90 mmHg or seated diastolic blood pressure (DBP) of <60 mmHg;
4. Patients with orthostatic hypotension;
5. Positive results of hepatitis B surface antigen, hepatitis C antibody, syphilis antibody and human immunodeficiency virus antibody.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of adverse event (AE), serious adverse event (SAE) | 7 days (SAD), 14 days (MAD)

SECONDARY OUTCOMES:
PK parameter of HRS-9813: Area under the concentration time curve (AUC) | Days 1-9
PK parameter of HRS-9813: Maximum Plasma Concentration (Cmax) | Days 1-9
PK parameter of HRS-9813: Time to maximum plasma concentration (Tmax) | Days 1-9
PK parameter of HRS-9813: Half-life (t1/2) | Days 1-9
PK parameter of HRS-9813: Apparent clearance (CL/F) | Days 1-9
PK parameter of HRS-9813: Apparent volume of distribution (Vz/F) | Days 1-9
PK parameter of HRS-9813: Accumulation ratio (Racc) | Days 1-9
PK parameter of HRS-9813: Cumulative amount excreted (Ae) in the urine | Days 1-2
PK parameter of HRS-9813: Fractional excretion (fe) in the urine | Days 1-2
PK parameter of HRS-9813: Renal clearance (CLR) | Days 1-2

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided